CLINICAL TRIAL: NCT05865652
Title: Evaluation of Membrane Phospholipid Metabolism and Cellular Energy Metabolism in Subjects at High Risk of Psychotic Transition
Brief Title: Evaluation of Membrane Phospholipid and Energy Metabolism in Subjects at High Risk of Psychotic Transition
Acronym: MR7T-UHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02708-33
Record Dates: First submitted 2022-04-21; First posted 2023-05-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Patients With Ultra High Risk of Psychotic Transition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Participants of this group are subjects with ultra high risk of psychotic transition.
  At inclusion visit, subjects will have a psychiatric evaluation and a cerebral MRI examination with phosphorus 31 Magnetic Resonance Spectroscopy in order to investigate membrane phospholipid metabolism and cellular energy metabolism.
  One and two years after the inclusion visit, subjects will have a psychiatric evaluation in order to objectivize if a psychotic transition has occured.
  Interventions: Diagnostic Test: Cerebral MRI with Phosphorus 31 Magnetic Resonance Spectroscopy
- Control group (Active Comparator): Participants of this group are healthy volunteers. Subjects will have one single visit with a psychiatric evaluation and a cerebral MRI examination with phosphorus 31 Magnetic Resonance Spectroscopy in order to investigate membrane phospholipid metabolism and cellular energy metabolism.
  Interventions: Diagnostic Test: Cerebral MRI with Phosphorus 31 Magnetic Resonance Spectroscopy

INTERVENTIONS:
Diagnostic Test: Cerebral MRI with Phosphorus 31 Magnetic Resonance Spectroscopy — Cerebral MRI with Phosphorus 31 Magnetic Resonance Spectroscopy

SUMMARY:
The management of schizophrenia is a major public health issue, due to its particularly disabling psychotic symptoms and their onset at an early age, typically in adolescents or young adults.

The physiopathological hypothesis of an anomaly relating to the renewal of cell membranes and energy metabolism in schizophrenia was proposed as early as the 1930s. This is based on anomalies at certain times in the development of the balance between phosphomonesters, precursors of membrane phospholipids, and phosphodiesters, catabolites of membrane phospholipids. Alterations of these different balances sign neurodevelopmental disorders, and can be objectified by specific techniques such as phosphorus-31 magnetic resonance spectroscopy (SMR-31P). This is used in particular to characterize the energy metabolism of the brain and allows in vivo quantification of phosphorus metabolites.

The application of SMR-31P techniques to assess the metabolism of membrane phospholipids and cellular energy metabolism in subjects at high risk of psychotic transition could make it possible to objectify a difference between subjects subsequently suffering from a psychotic transition compared to those who do not suffer from it. Alterations in the metabolism of membrane phospholipids could thus represent a biomarker of psychotic transition. Secondarily, this approach would make it possible to provide elements as to the validity as a diagnosis of this category, which is very heterogeneous in its future.

Among the Ultra High Risk (UHR) group, subjects with a psychotic transition (UHR-T) are compared to subjects without this transition (UHR-NT) during the two years of follow-up.

The UHR group is compared to the control group.

At T0, UHR patients and healthy volunteers will perform brain MRI with Phosphorus 31 magnetic resonance spectroscopy.

UHR patients will then be reviewed:

* at T+1 year for a clinical assessment medical interview to assess the patient's functioning and the appearance of symptoms;
* at T+2 years for the realization of a follow-up interview with passing of the scales CAARMS (Comprehensive Assessment of At Risk Mental State) and SOFAS (scale of evaluation of the social and professional functioning) in order to determine if the subject belongs to the UHR-T or UHR-NT group.

ELIGIBILITY:
Inclusion Criteria for the UHR group:

* Patient between 15 and 25 years old
* Patient fulfilling the UHR criteria objectified by the Comprehensive Assessment of At Risk Mental State scale (CAARMS) and by the social and professional functioning assessment scale (SOFAS) (the "Vulnerability" group is also taken into account, combining first-degree history and functional impact.)
* Patient with no contraindication to performing a 7T MRI examination
* Affiliated patient or beneficiary of a social security scheme.
* Free, informed consent, written and signed by the participant, the investigator and the legal representative if applicable (at the latest on the day of inclusion and before any examination required by the research).

Inclusion Criteria for the Control group:

* Subjects aged 15 to 25 years old,
* healthy volunteer subject or subject to benefit from an imaging examination, not presenting the criteria of a mental health disorder objectified by a medical interview
* Subject with no contraindication to performing a 7T MRI examination
* Affiliated subject or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant, the investigator and the legal representative if applicable (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria for the UHR group:

* Patient not at risk or already in a psychotic pathological process according to DSM-5 criteria.
* Patient already receiving antipsychotic treatment or whose background treatment was changed less than a month ago.
* Patient presenting an absolute contraindication to 7T MRI such as: foreign bodies (intracranial clips, vascular magnetic clips, cardiac or neural pacemakers, stents, coils, implantable chamber, intracorporeal metallic splinters, cochlear implants, intracorporeal metallic foreign bodies, mechanical heart valve, implanted injection pump, non-removable piercings), pregnant woman, allergy to contrast products, moderate to severe renal insufficiency, breastfeeding, implanted contraception, tinnitus, claustrophobia and braces.

The relative contraindications are to be considered, namely: previous surgical interventions, medically implanted device, tattoo or permanent make-up.

Exclusion criteria for the control group:

- Subject presenting an absolute contraindication to 7T MRI such as: foreign bodies (intracranial clips, vascular magnetic clips, cardiac or neural pacemakers, stents, coils, implantable chamber, intracorporeal metallic fragments, cochlear implants, intracorporeal metallic foreign bodies, valve mechanical heart, implanted injection pump, non-removable piercings), pregnant woman, allergy to contrast products, moderate to severe renal insufficiency, breast-feeding, implanted contraception, tinnitus, claustrophobia and braces.

The relative contraindications are to be considered, namely: previous surgical interventions, medically implanted device, tattoo or permanent make-up.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Difference of cellular inorganic phosphate between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of inorganic phosphate.
Difference of cellular phosphocreatine between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of phosphocreatine.
Difference of cellular Gamma ATP between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of Gamma ATP.
Difference of cellular Alpha ATP between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of Alpha ATP.
Difference of cellular beta ATP between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of beta ATP.
Difference of intracellular pH between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of intracellular pH.
Difference of membrane phosphodiester alterations between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of phosphodiester.
Difference of membrane phosphomonoester alterations between UHR-T and UHR-NT patients. | 2 years
  Levels measurements of phosphomonoester.

SECONDARY OUTCOMES:
Difference of cellular inorganic phosphate between UHR subjects and control subjects. | 2 years
  Levels measurements of inorganic phosphate.
Difference of cellular phosphocreatine between UHR subjects and control subjects. | 2 years
  Levels measurements of phosphocreatine.
Difference of cellular Gamma ATP between UHR subjects and control subjects. | 2 years
  Levels measurements of Gamma ATP.
Difference of cellular Alpha ATP between UHR subjects and control subjects. | 2 years
  Levels measurements of Alpha ATP.
Difference of cellular beta ATP between UHR subjects and control subjects. | 2 years
  Levels measurements of beta ATP.
Difference of cellular intracellular pH between UHR subjects and control subjects. | 2 years
  Levels measurements of intracellular pH.
Difference of membrane phosphodiester alterations between UHR subjects and control subjects. | 2 years
  Levels measurements of phosphodiester.
Difference of membrane phosphomonoester alterations between UHR subjects and control subjects. | 2 years
  Levels measurements of phosphomonoester.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No